CLINICAL TRIAL: NCT06756568
Title: The Diagnostic Utility of Ultrasound in Pelvic Inflammatory Disease (PID)
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/037
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Pelvic Inflammatory Disease
MeSH Terms: conditions — Pelvic Inflammatory Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Reduced Morbidity — Early and accurate diagnosis using ultrasound minimizes delays in treatment initiation, thereby preventing complications such as chronic pain and abscess formation. By reducing the severity and duration of the disease, ultrasound contributes to improved patient well-being and a quicker recovery trajectory.

SUMMARY:
Pelvic inflammatory disease (PID) represents a significant and complex health issue affecting women, particularly those of reproductive age. Characterized by the infection and inflammation of the reproductive organs, PID often results from ascending infections primarily caused by sexually transmitted pathogens, such as Neisseria gonorrhoeae and Chlamydia trachomation. However, it can also be associated with endogenous bacteria or occur following surgical procedures.

DETAILED DESCRIPTION:
The diverse manifestations of PID from asymptomatic cases to acute presentations, pose significant challenges in diagnosis and prompt treatment. Accurate diagnosis is crucial, as untreated infections can lead to severe complications, including infertility, chronic pelvic pain, and ectopic pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age (18-45 years) presenting with symptoms suggestive of pelvic inflammatory disease (PID).
* Patients who have been clinically diagnosed with PID based on symptoms such as lower abdominal pain, fever, abnormal vaginal discharge, and tenderness upon pelvic examination.
* Patients who have undergone preliminary diagnostic tests, such as high vaginal swab (HVS) and urine microscopy, culture, and sensitivity (m/c/s), prior to ultrasound assessment.

Exclusion Criteria:

* Pregnant women, due to potential confounding factors in ultrasound findings and differential diagnosis.
* Patients with chronic pelvic pain not related to acute PID episodes.
* Patients who do not provide informed consent for participation in the study.
* Patients with a history of recent pelvic surgery within the last 6 months, as postoperative changes may affect ultrasound findings.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pelvic Inflammatory Disease
Study Population: to check the Pelvic Inflammatory Disease (PID) using Ultrasound
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2024-02-18 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-02-16 (Estimated)

PRIMARY OUTCOMES:
ultrasound | 12 Months
  Ultrasound (GE Logiq P7 convex probe.3.5-5MHz) imaging using a curvilinear transducer that provides a broad field of view, commonly used for evaluating abdominal and pelvic organs.
  Doppler flow characteristics which increased blood flow in the pelvic region, especially around the fallopian tubes or ovaries, as detected by color Doppler ultrasound, indicative of inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- Lady Reading Hospital, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No